CLINICAL TRIAL: NCT06122012
Title: A Study to Evaluate the Efficacy and Safety of HSK16149 Capsule Combined With L-carnitine Hydrochloride Tablets and Lipoic Acid Combined With L-carnitine Hydrochloride Tablets in Diabetic Peripheral Neuralgia Patients in China
Brief Title: To Evaluate the Efficacy and Safety of HSK16149 With L-carnitine in Diabetic Peripheral Neuralgia Patients in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK16149-206
Record Dates: First submitted 2023-10-25; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — BID protein, human; Thioctic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK16149 capsule combined with L-carnitine hydrochloride (Other): HSK16149 capsule (20 mg/ capsule) was administered orally, 1 capsule twice a day for 12 weeks. Acetyl-l-carnitine hydrochloride tablets (0.25g/ tablet) were administered orally after meals, 2 tablets 3 times a day for 12 weeks
  Interventions: Drug: HSK16149 20mg BID
- Lipoic acid combined with L-carnitine hydrochloride (Other): HSK16149 capsule (20 mg/ capsule) was administered orally, 1 capsule twice a day for 12 weeks. Lipoic acid tablets (0.3g/ tablet) were administered half an hour before breakfast, 2 tablets once a day for 11 weeks.
  Interventions: Drug: HSK16149 20mg BID

INTERVENTIONS:
Drug: HSK16149 20mg BID — HSK16149 20mg BID with L-carnitine hydrochloride tablets 2 tablets TID ；Lipoic acid tablets 2 tablets BID with L-carnitine hydrochloride tablets 2 tablets TID；
  Other Names: Lipoic acid tablets 2 tablets BID；L-carnitine hydrochloride tablets 2 tablets TID

SUMMARY:
Observe the effects of HSK16149 capsule combined with acetyl-L-carnitine hydrochloride tablets and lipoic acid combined with acetyl-L-carnitine hydrochloride tablets Efficacy and safety in diabetic peripheral neuralgia patients in China

DETAILED DESCRIPTION:
Observe the effects of HSK16149 capsule combined with acetyl-L-carnitine hydrochloride tablets and lipoic acid combined with acetyl-L-carnitine hydrochloride tablets Efficacy and safety in diabetic peripheral neuralgia patients in China.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign written informed consent;
2. Male or female over the age of 18 (including the threshold);
3. Diabetic peripheral neuralgia (DPNP) diagnosis;
4. The average pain Visual Analogue Scale (VAS) score in the past 24 h was assessed as ≥ 40 mm and < 90 mm during screening.

Exclusion Criteria:

* 1. Peripheral neuropathy or pain unrelated to DPN that the investigator determined might confuse the DPNP assessment;

  2. History of malignant tumors (excluding cured basal cell carcinoma of the skin, carcinoma in situ, and papillary thyroid carcinoma) or history of antitumor therapy within 5 years prior to screening;

  3. Severe abnormal liver and kidney function, meeting any of the following clinical laboratory test results:
  1. Liver function: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × upper limit of normal (ULN); Or total bilirubin (TBIL) > 1.5 × ULN;
  2. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 (calculated according to simplified MDRD formula);

  4. Known allergic history to test drug components or other drugs or excipients with similar chemical structure;

  5. Past suicidal behavior or suicidal intention;

  6. Women who are pregnant, planning to become pregnant during the study period, or breastfeeding; Women who do not wish to use reliable contraceptive methods (including condoms, spermicides, or Iuds) for 28 days after signing up for the ICF from the beginning to the last trial drug administration, or who plan to use progesterone contraceptives during this period;

  7. Participated in any other clinical studies within 30 days prior to screening;

  8. The researcher determines that there are other conditions that are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy and safety of HSK16149 capsule combined with acetyl-L-carnitine hydrochloride tablet and lipoic acid combined with acetyl-L-carnitine hydrochloride tablet in the treatment of diabetic peripheral neuralgia | week12
  Using the Analysis of Covariance (ANCOVA) model, changes in ADPS relative to baseline at 12 weeks of treatment were taken as dependent variables, and baseline values of study centers, groups, and ADPS were taken as explanatory variables, and the adjusted least squares mean and standard errors of each group were listed. The difference and 95% confidence interval of the mean change of ADPS from baseline at 12 weeks in the HSK16149 capsule combined with acetyl-L-carnitine hydrochloride group compared with the lipoic acid combined with acetyl-L-carnitine hydrochloride group were calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China